CLINICAL TRIAL: NCT00442026
Title: A Multicenter Randomized Phase III Study of the Docetaxel and Gemcitabine Combination Versus Monotherapy With Gemcitabine as First-line Treatment in Elderly Patients With Advanced Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: Randomized Trial of Docetaxel and Gemcitabine Versus Gemcitabine in Elderly Patients With NSCLC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/06.11
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Cancer; NSCLC; Elderly; Chemotherapy; Docetaxel; Gemcitabine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): DG
  Interventions: Drug: Docetaxel; Drug: Gemcitabine
- 2 (Experimental): G
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Docetaxel — Docetaxel at the dose of 30mg/m2 IV on days 1 and 8 every 3 weeks for 6 consecutive cycles
  Other Names: Taxotere
  Arms: 1
Drug: Gemcitabine — Gemcitabine at the dose of 900mg/m2 IV on days 1 and 8 every 3 weeks for 6 consecutive cycles
  Other Names: Gemzar
  Arms: 1
Drug: Gemcitabine — Gemcitabine at the dose of 1200mg/m2 IV on days 1 and 8 every 3 weeks for 6 consecutive cycles
  Other Names: Gemzar
  Arms: 2

SUMMARY:
This trial will compare the efficacy of the docetaxel and gemcitabine combination versus monotherapy with gemcitabine as first-line treatment in elderly patients with advanced NSCLC

DETAILED DESCRIPTION:
Docetaxel and gemcitabine are well known active agents in the treatment of NSCLC. The standard treatment of elderly patients with advanced NSCLC is monotherapy with a third generation agent. However, there are only few randomized trials evaluating a two drug combination specifically addressed to elderly patients. The role of comprehensive geriatric assessment in treatment efficacy and tolerance is an area of investigation

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically- confirmed Non-Small-Cell Lung Cancer
* Stage IIIB/IV
* No prior chemotherapy
* Presence of two-dimensional measurable disease. The measurable disease should not have been irradiated.
* Absence or irradiated and stable central nervous system metastatic disease
* Life expectancy of more than 3 months
* Age ≥ 70 years.
* Performance status (WHO) < 3
* Patients "non-frail" according to comprehensive geriatric assessment
* Adequate bone marrow function (Absolute neutrophil count > 1000/mm^3, Platelet count > 100000/mm^3, Hemoglobin > 9gr/mm^3).
* Adequate liver (Bilirubin < 1.5 times upper limit of normal and SGOT/SGPT < 2 times upper limit of normal) and renal function (creatinine < 2mg/dl).
* Adequate cardiac function (LVEF > 50%).
* Informed consent.

Exclusion Criteria:

* Psychiatric illness or social situation that would preclude study compliance.
* Other concurrent uncontrolled illness.
* Other invasive malignancy within the past 5 years except nonmelanoma skin cancer.
* No presence of a reliable care giver
* Other concurrent investigational agents.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Overall survival between the two treatment arms | Probability of 1 year survival (%)

SECONDARY OUTCOMES:
Overall response rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)
Time to disease progression | 1 year
Quality of life assessment | Assessment every two cycles
Toxicity profile | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Lampros Vamvakas, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology; Athanasios Karampeazis, MD, Principal Investigator — University Hospital of Crete
Locations (9):
- Greece (9):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital, Medical Oncology Unit, Athens
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - Sismanogleio General Hospital, 1st, 2nd Dep of Pulmonary Diseases, Athens
  - Sotiria" General Hospital, 1st, 3rd, 8th Dep of Pulmonary Diseases, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus,1st Dep of Medical Oncology, Piraeus
  - Theagenion" Anticancer Hospital of Thessaloniki, Thessaloniki

REFERENCES:
- [Derived] Karampeazis A, Vamvakas L, Kotsakis A, Christophyllakis C, Kentepozidis N, Chandrinos V, Agelidou A, Polyzos A, Tsiafaki X, Hatzidaki D, Georgoulias V. Docetaxel plus gemcitabine versus gemcitabine in elderly patients with advanced non-small cell lung cancer and use of a geriatric assessment: Lessons from a prematurely closed Hellenic Oncology Research Group randomized phase III study. J Geriatr Oncol. 2017 Jan;8(1):23-30. doi: 10.1016/j.jgo.2016.05.002. Epub 2016 Jun 2. PMID 27264267